CLINICAL TRIAL: NCT01507844
Title: Continuous Positive Airway Pressure Effect on Air Trapping, Endurance Time in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Continuous Positive Airway Pressure Effect on Air Trapping in Chronic Obstructive Pulmonary Disease Patients
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 86/09; 12 (Other: Israel lung Association)
Record Dates: First submitted 2009-11-02; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; CPAP; Sham; FEV1; IC; RV/TLC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- ventilation (Sham Comparator)
  Interventions: Device: positive ventilation

INTERVENTIONS:
Device: positive ventilation — 10 minutes of increased 4,7,12 positive pressure ventilation
  Other Names: CPAP

SUMMARY:
Chronic obstructive pulmonary disease is a disease characterized by small airways inflammation and obstruction. The small airways disease produces hyperinflation (air trapping), which increases with exercise. Continuous positive airways pressure may reduce small airways obstruction and therefore air trapping. Pulmonary function tests including lung volumes at rest and and after exercise will be measured. In addition, exercise endurance time before treatment and after treatment will be measured.

DETAILED DESCRIPTION:
Continuous positive airways pressure which prevent small air ways collapse and may also clear secretions. At first stage the optimal pressure for reducing air trapping will be determined. In addition, all patients will undergo a maximal exercise test. A baseline complete pulmonary function test is performed followed by continuous positive air way pressure at the pre-determined pressure. This will be followed by exercise at 60% of maximal obtained previously.

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive lung disease stage 2-3 GOLD
* FRC > 120%

Exclusion Criteria:

* active ischemic heart disease
* heart failure
* peripheral vascular disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
improved small airways obstruction | 2-3 hrs
  Following CPAP ventilation measurement be repeated for 3 hrs

SECONDARY OUTCOMES:
improved respiratory symptoms | 2-3 hrs
  CAT score

CONTACTS AND LOCATIONS:
Overall Officials: David stav, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Pulmonary Institute, Beer Yaakov, Israel